CLINICAL TRIAL: NCT01465529
Title: A Double-blind, Randomized, Placebo-controlled, Cross-over Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of Alginate Oligosaccharide (OligoG) Administered for 28 Days in Subjects With Cystic Fibrosis Chronically Colonised With Pseudomonas Aeruginosa
Brief Title: A Cross-over Study of OligoG in Subjects With Cystic Fibrosis. Fibrosis
Acronym: OligoG
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AlgiPharma AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMR-2375; 2010-023090-19 (EudraCT Number)
Record Dates: First submitted 2011-10-31; First posted 2011-11-04 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — oligoG CF-5-20; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental)
  Interventions: Drug: OligoG CF-5/20
- Placebo (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: OligoG CF-5/20 — 6% OligoG CF-5/20 in water
  Other Names: OligoG
  Arms: Active
Drug: Saline — 0.9% NaCl in water
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and local tolerability of multiple dose administration of inhaled OligoG in CF subjects. Particular emphasis will be put on local, clinical tolerance, pulmonary function and pulmonary adverse events. The secondary purpose is to monitor the effect of multiple dose administration of inhaled OligoG on various efficacy variables, such as mucolytic activity, lung function, respiratory symptoms, Quality-of-Life and microbiological outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with a confirmed diagnosis of cystic fibrosis defined by:

  * Clinical features consistent with the diagnosis of CF [(Rosenstein BJ and Cutting GR 1998)]; AND
  * Sweat chloride ≥60 mmol/L by pilocarpine iontophoresis; OR
  * Genotypic confirmation of CFTR mutation
* Aged 18 years or older
* Ability to provide samples for microbiological evaluation throughout the study. Note: sputum samples are preferred however cough swabs may be performed on occasions where sputum cannot be collected.
* Positive microbiological finding of Pseudomonas aeruginosa in expectorated sputum or cough swab documented within 24 months prior to Screening (Visit 1).
* FEV1 must, at Screening (Visit 1), be between 35%-80% of the predicted normal value following adjustment for age, gender, and height according to the Knudson equation [(Knudson RJ., Lebowitz MD., et al 1983)].
* At Screening (Visit 1), no clinical or laboratory findings suggestive of significant pulmonary illness, other than CF, which in the opinion of the investigator would preclude participation in the study.
* Female subjects of child bearing potential and male subjects participating in the study who are sexually active must use acceptable contraception. Female subjects documented as being of non child-bearing potential (Section 4.2.8) are exempt from the contraceptive requirements. For the purpose of this study acceptable contraception is defined as:

  * oral, injected or implanted hormonal methods of contraception;OR
  * placement of an intrauterine device (IUD) or intrauterine system (IUS);OR
  * barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository
* Provision written informed consent

Exclusion Criteria:

* Changes in underlying therapy (e.g., pulmonary massage therapy, bronchodilators, NSAIDs, antibiotic agents, pancreatic enzyme preparations, nutritional supplements and DNase within the 21 days prior to Day 1 (Visit 2). Subjects must be willing to remain on the same underlying stable therapy regimens for the duration of the study until the final follow-up visit at Day 111.
* Changes in physiotherapy technique or schedule within 14 days prior to Day 1 (Visit 2).
* Prohibited medications within 7 days prior to Day 1 (Visit 2). Prohibited medications are described in Section 5.6
* Pulmonary exacerbation within 28 days of Screening (Visit 1).
* Positive microbiological finding of Burkholderia sp. in expectorated sputum or cough swab documented within 12 months prior to Screening (Visit 1).
* On-going acute illness. Subjects must not have needed an outpatient visit, hospitalization or required any change in therapy for other pulmonary disease between Screening (Visit 1) and Day 1 (Visit 2).
* History of, or planned organ transplantation.
* Allergic bronchopulmonary aspergillosis (ABPA) in the last 12 months prior to Screening (Visit 1), defined as having received treatment for ABPA.
* Requirement for continuous (24 hour/day) oxygen supplementation.
* Concomitant administration of inhaled mannitol or hypertonic saline within 7 days prior to Day 1 (Visit 2).
* Initiation of cycled, inhaled tobramycin (TOBI) less than 4 months prior to Screening (Visit 1). Note: Chronic TOBI users are allowed to participate in this study, but subjects who have recently initiated chronic TOBI should have at least 2 cycles of TOBI in the preceding 4 months before being enrolled in this study. Chronic TOBI subjects should be starting an 'off- TOBI' period at Day 1 (Visit 2) so there will be no concomitant dosing of TOBI and assigned study medication.
* Clinically significant abnormal findings on haematology or clinical chemistry. In addition, any value ≥ 3 x the upper limit of normal will exclude the subject from participating in the study.
* Subjects unable to perform pulmonary function tests according to the ATS/ERS criteria.
* Pregnant or breast-feeding women. A negative urine pregnancy test must be demonstrated in females of child-bearing potential (Section 4.2.8) at Screening (Visit 1).
* Subjects who have participated in any interventional clinical trial within the 28 days prior to Day 1 (Visit 2).
* Subjects with documented or suspected, clinically significant, alcohol or drug abuse. The determination of clinical significance will be determined by the Investigator.
* Known allergies or intolerance to alginates (e.g., foods and food additives based on seaweed extracts).
* Current malignant disease (with the exception of basal cell carcinoma; BCC).
* Any serious or active medical or psychiatric illness, which in the opinion of the Investigator, would interfere with subject treatment, assessment, or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-05; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Safety and local tolerability of multiple dose administration of inhaled OligoG in Cystic Fibrosis subjects. | Day 111 + 6 month follow-up

SECONDARY OUTCOMES:
The effect of multiple dose administration of inhaled OligoG on various efficacy variables | Day 111 + 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Martin Walshaw, MD, Principal Investigator — Liverpool Heart & Chest Hospital, UK
Locations (3):
- Ireland (2):
  - Beaumont Hospital, Dublin
  - University College Hospital Galway, Galway
- Liverpool Heart & Chest Hospital, Liverpool, United Kingdom